CLINICAL TRIAL: NCT00003715
Title: A Prospective, Randomized, Open-Label, Comparative Clinical Trial in Post-Surgical Melanoma Patients With Either DNP-Modified Autologous Tumor Vaccine or Interferon Alpha-2b
Brief Title: Vaccine Therapy Compared With Interferon Alfa in Treating Patients With Stage III Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated: recruiting or enrolling participants has halted prematurely and will not resume; participants are no longer being examined or treated
Sponsor: AVAX Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066824; AVAX-A/100/0101
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — BCG Vaccine; FANG vaccine; Interferon-alpha; Drug Therapy; Cyclophosphamide

INTERVENTIONS:
Biological: BCG vaccine
Biological: autologous tumor cell vaccine
Biological: recombinant interferon alfa
Drug: chemotherapy
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Vaccines made from a person's melanoma cells may make the body build an immune response to kill tumor cells. Interferon alfa may interfere with the growth of the cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of melanoma vaccine with that of interferon alfa-2b in treating patients who have stage III melanoma that has spread to regional lymph nodes following surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the relapse-free and overall survival rates in patients with stage III melanoma treated with autologous tumor vaccine versus interferon alfa-2b as postsurgical adjuvant therapy. II. Compare the safety and tolerability of these regimens in this patient population.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to number of metastatic lymph node sites (1 vs more than 1), number of positive lymph nodes in a single site (none vs 1 or more), presence of intransit metastases (yes vs no), and evidence of extranodal extension (yes vs no). Patients are randomized to one of two treatment arms. Arm I: Patients receive autologous tumor cell vaccine intradermally once a week for 7 weeks followed by a booster injection at 6 months. BCG is given concurrently with vaccine as an immune-stimulator for doses 2-8. Patients also receive cyclophosphamide 6 days after the first vaccine injection. Arm II: Patients receive interferon alfa-2b IV for 5 consecutive days a week for 4 weeks followed by maintenance doses given subcutaneously 3 times a week for 48 weeks. Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 386-425 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed melanoma metastatic to regional lymph nodes with a clinically palpable mass Must have clinical evidence of the following: Metastases in 1 nodal site All other nodes microscopically negative No intransit metastases No extranodal extension OR Metastases in more than 1 nodal site More than 1 positive lymph node in a single site Intransit metastases Extranodal extension Must have undergone complete resection of tumor, measuring at least 2 cm in diameter, within the past 6 weeks No distant metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 80-100% Life expectancy: At least 6 months Hematopoietic: Hematocrit at least 30% WBC at least 3,000/mm3 Hepatic: Hepatitis B and C negative Renal: Not specified Other: Not pregnant or nursing No active serious infection No active autoimmune disease HIV negative No other malignancy within the last 5 years except squamous cell carcinoma of the skin, carcinoma in situ of the cervix, superficial bladder carcinoma, early stage prostate cancer, or noninvasive melanoma No active severe depression or psychiatric disorder with psychotic symptoms No uncontrolled thyroid abnormalities

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 weeks since prior cytotoxic drugs (except for isolated limb perfusion) Endocrine therapy: No concurrent systemic corticosteroids Radiotherapy: At least 6 months since prior radiotherapy Surgery: See Disease Characteristics Other: At least 30 days since prior investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Karen Doak, Study Chair — AVAX Technologies
Locations (17):
- United States (17):
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Columbia - HCA Cancer Research Network, North Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Georgia Cancer Specialists, Decatur, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - Midwest Oncology Consortium, Kansas City, Missouri
  - Jersey Shore Cancer Center, Neptune City, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Palmetto Hematology/Oncology Associates, Spartanburg, South Carolina